CLINICAL TRIAL: NCT00951145
Title: Medium and Long Term Outcome of Total Hip Arthroplasty Using Accolade TMZF Femoral Stem
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Javad Parvizi, MD, FRCS, Rothman Institute
Other Study IDs: RIFJPAR 09-01
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Osteoarthritis of the Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective/prospective study evaluating the clinical and radiographic outcome of total hip arthroplasty (THA) performed using Accolade femoral stem in a consecutive group of patients. All patients eligible for inclusion will be identified. The investigators hypothesize that the outcome of THA performed using Accolade femoral stem is equal or superior to historical survivorship of THA using other types of collarless, proximally coated, tapered stems.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing THA prior to 1/1/2003 using Accolade femoral stem.
2. Patients with hip fracture undergoing THA will also be included.
3. Patients willing and able to comply with follow-up requirements and self-evaluations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing THA prior to 1/1/2003 using Accolade femoral stem
Sampling Method: Probability Sample

PRIMARY OUTCOMES:
The outcome of THA performed using Accolade femoral stem is equal or superior to historical survivorship of THA using other types of collarless, proximally coated, tapered stem

SECONDARY OUTCOMES:
Proximally coated tapered stems can be used for patients with various bone types, bone morphology, and underlying diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Parvizi Javad, MD, Principal Investigator — Rothman Institute; Hozack William, MD, Principal Investigator — Rothman Institute
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States